CLINICAL TRIAL: NCT04129463
Title: SST With Iris Incarceration in Buphthalmous
Brief Title: Subscleral Trabeculectomy With Iris Incarceration in Buphthalmous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaaban Elwan (Other)
Responsible Party: Sponsor-Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minia University, SST
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Iris Incarceration
Keywords: Buphthalmous; Iris incarceration; SST; IOP; AXL

STUDY DESIGN:
Intervention Model Description: Group 1 SST with iris incarceration and group2 conventional trabeculotomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SST with Iris incarceration (Active Comparator): infants that underwent SST with iris incarceration procedure
  Interventions: Device: Subscleral Trabeculectomy (SST) with Iris incarceration
- Conventional trabeculotomy (Active Comparator): infants that underwent Conventional trabeculotomy
  Interventions: Device: Conventional trabeculotomy

INTERVENTIONS:
Device: Subscleral Trabeculectomy (SST) with Iris incarceration — Subscleral Trabeculectomy with Iris Incarceration using iris forceps and scissors
  Other Names: Group1
  Arms: SST with Iris incarceration
Device: Conventional trabeculotomy — Conventional trabeculotomy in Buphthalmous using rigid Hans trabeculotome
  Other Names: Group 2
  Arms: Conventional trabeculotomy

SUMMARY:
Purpose: To evaluate a new modification for surgical treatment of Buphthalmous using subscleral trabeculectomy (SST) with iris incarceration Design: Prospective, randomized, consecutive interventional comparative study. Setting: Ophthalmology department, Faculty of Medicine, Minia University, 61519, El-Minia, Egypt.

Patients and Methods:

This was a prospective study of eyes of 40 eyes with buphthalmous in 25 child 15 bilateral and 10 with unilateral Buphthalmous divided into 2 groups. Group 1 (20 eyes ) those underwent subscleral trabeculectomy (SST) with iris incarceration a new modification to SST and group 2 conventional rigid trabeculotomy through a period of 4 years between Jan., 2015 and Feb., 2019. Patient's data of 2 years follow-up were recorded. The primary outcomes were the mean intraocular pressure (IOP) control in which complete success was defined as an IOP ≤18 mm Hg without the use of anti-glaucoma drugs and a qualified success when medications were used to reach this target and times of another surgical interference till reach IOP control. The secondary outcomes were studding bleb formation, the change in corneal diameter (CD), cup disc ratio (C/D) , and axial length (AXL)

DETAILED DESCRIPTION:
Subjects and Methods This was a prospective study of eyes of 40 eyes with Buphthalmous in 25 infants (15 bilateral and 10 with unilateral) divided into 2 groups. Group 1 (20 eyes) those underwent Subscleral trabeculectomy (SST) with iris incarceration a new modification to SST and group 2 conventional rigid trabeculotomy through a period of 4 years between Jan., 2015 and Feb., 2019. The local board committee approved the study as well as all patients' relatives signed consent and the study was in agreement with Declaration of Helsinki Tents. The primary outcomes were the mean intraocular pressure (IOP) measured under General Anesthesia (GA) and the number of repeated surgical intervention. Complete success was defined as an IOP ≤18 mm Hg without the use of anti-glaucoma drugs, a qualified success when medications were used to reach this target and failure if the target IOP would not be reached in spite of full anti-glaucoma medication and the infant needs another anti-glaucoma procedure and the number of repeated surgical intervention were recorded. The secondary outcomes were studding bleb formation, the change in corneal diameter (CD), cup disc ratio (C/D), and axial length (AXL).

Preoperative examinations: History taking including, age, sex, laterality, family history and consanguinity, anti-glaucoma drugs. Ophthalmological examinations were done under GA, includes slit lamp examination, corneal clarity, horizontal corneal diameter, fundus examination and measurement of cup disc ratio, IOP with Perkins tonometer, and axial length by ultrasonography. The demographic data were registered as in (Table 1).

Surgical procedure:

All procedures were done by one of the Authors under GA. In group 1 SST with iris incarceration Steps in brief:-

* Clear corneal traction suture by vicryl 7/0 in the superior peripheral part 1 mm from the limbus
* Conjunctival peritomy with fornix based conjunctival flap was done in the upper temporal quadrant.
* Half thickness rectangular scleral flab 3.5 x 4.5 mm was constructed.
* Paracentesis to lower IOP and allows reformation of anterior chamber when needed and check filtration.
* Block trabeculectomy were done manually by knife and vannas scissors.
* Iris incarceration was done by cutting the iris into 2 pillars, one pillar incarcerated under the scleral flap and the other one reposted with iris repositor resulting in inverted coma shaped pupil.
* Scleral flap was closed with interrupted 10/0 nylon suture and Conjunctival flap with contentious 10/0 nylon suture then injection of subconjunctival steroid, antibiotic and eye dressing.

In group 2 trabeculotomy Steps in brief:-

* Conjunctival peritomy with fornix based Conjunctival flap was done in the upper temporal quadrant.
* Superficial rectangular scleral flab 3.5 x 4.5 mm and then small triangular deep scleral flab (modified technique) with deroofing of Schlemm's canal anteriorly to the scleral spur were done.
* Radial incision into the scleral bed and cutting Schlemm's canal, exposure of its opening and dilatation of the ostia by injection of Healon or trabeculotome.
* Paracentesis to lower IOP allows reformation of anterior chamber when needed and check filtration.
* Hans's trabeculotome was inserted into Schlemm's canal from one side and centripetal rupture of the canal through trabecular meshwork into the anterior chamber about 70- 90 degree and repeated on the other side.
* Scleral flap was closed with interrupted 10/0 nylon suture and Conjunctival flap with contentious 10/0 nylon suture then injection of subconjunctival steroid, antibiotic and eye dressing

Post-operative management:

The patients were prescribed topical tobradex (tobramycin- dexamethasone) eye drops QID and tapering through 4-6 weeks and Vigamox (moxifloxacin 0.3 mg, Alcon Co) eye drops QID for 2 weeks. Scheduled follow up visits were advised next postoperative day, one week, monthly for three months then each three months for 2 years. Each visit the child subjected to full ophthalmological examinations previously mentioned and antiglaucoma medications were prescribed when needed (IOP>18 mmHg) or glaucoma progression starting by one drug beta blockers and adding dorzolamide or prostaglandin to reach the target IOP. Another glaucoma procedure were done if the IOP > 18 mmHg with maximum tolerated medication. Patient's data of the 2 years follow-up were recorded. The results of one week, 1 month, 3 months, 6 months, 1 year and 2 years were included in the statistical analysis.

Statistical analysis:

Data were collected, for statistical analysis done by using SPSS statistical package version 20. Descriptive statistics for the (mean ±SD) were done. Paired student's t-test was used for comparison of two related parameters preoperative and postoperative. For all tests (P value) was considered significant if < 0.05.

ELIGIBILITY:
Inclusion Criteria:

The study included infants aged below ≤ 1 year with Buphthalmous with or without antiglaucoma medications and not had previous antiglaucoma surgery.

-

Exclusion Criteria:

* Eyes that had previous antiglaucoma procedure or eyes that need combined operation and infants not fit for GA.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
IOP reduction | 2 years
  Intra-ocular pressure change in mmHg

SECONDARY OUTCOMES:
Corneal diameter | 2 years
  Corneal diameter change in mm
Cup/ disc change | 2 years
  Cup/ disc change in mm
AXL change | 2 years
  Axial length change in mm

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban AM Elwan, MD, Principal Investigator — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data share
Supporting Information: CSR
Time Frame: 2 years
Access Criteria: Data